CLINICAL TRIAL: NCT03793985
Title: Phase I Clinical Trial to Compare the Pharmacokinetics and Safety of CKD-391 With Co-administration of D086 and D337 in Healthy Adult Volunteers
Brief Title: Compare the Pharmacokinetics and Safety of CKD-391 With Co-administration of D086 and D337
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 152BE17006
Record Dates: First submitted 2018-12-13; First posted 2019-01-04 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (R+T+R+T) (Experimental): Period 1 : R Period 2 : T Period 3 : R Period 4 : T
  Interventions: Drug: T; Drug: R
- B (T+R+T+R) (Active Comparator): Period 1 : T Period 2 : R Period 3 : T Period 4 : R
  Interventions: Drug: T; Drug: R

INTERVENTIONS:
Drug: T — CKD-391 40/10mg
  Other Names: Test Drug
Drug: R — D086 and D337 co-administration
  Other Names: Reference drug

SUMMARY:
Compare the pharmacokinetic characteristics and safety between CKD-391 tablet and D337, D337 combination

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 aged and 45 aged in healthy male adult
2. Over 50 kg, BMI between 18.0-29.0 kg/m2
3. Subjects in good health as determined by physical exams and medical examinations. No congenital or chronic diseases and no abnormal signs determined by medical examinations.
4. Not abnormal or not clinically significant lab values.
5. Subjects who signed informed consent form with good understandings after explanations by investigators.

Exclusion Criteria:

1. No history or presence of clinically significant diseases.
2. Subjects showing adverse reaction to investigational product
3. Genetic problems in galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption.
4. History of myopathy
5. Subjects with abnormal lab values at least one below 1) AST or ALT>2 fold of upper normal limit 2) Total bilirubin>2 fold of upper normal limit 3) CK>2 fold of upper normal limit 4) Estimated Glomerular filtration rate<60mL/min/1.73m2
6. Drink over 21 units/week (1 unit= 10g=12.5mL of pure alcohol) or unable to stop drinking during clinical trials
7. Smoke over 10 cigarettes per day or unable to stop smoking
8. Subjects who previously participated in other clinical trials within 90 days
9. Subjects who donated whole blood within 60 days or donated component blood within 30 days or received blood transfusion within 30 days
10. Subjects who took any prescribed medications or oriental medicines within 14 days, or took any pharmacy medicines within 10 days.
11. Taking medications which induce or block medication metabolism
12. History of drug abuse
13. Subjects who took any prescribed medications or oriental medicines within 14 days, or took any pharmacy medicines within 7 days.
14. Disagree to contraception
15. Subjects who are in any conditions impossible participating in the clinical trials

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Cmax | 0~72hours
  To evaluate pharmacokinetic equivalence of experimental arm comparing Cmax
AUCt | 0~72hours
  To evaluate pharmacokinetic equivalence of experimental arm comparing AUCt

CONTACTS AND LOCATIONS:
Locations (1):
- INHA University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No